CLINICAL TRIAL: NCT01400958
Title: A Randomized, Double Blind, Placebo-Controlled Study Evaluating the Effect of Nuvigil® (Armodafinil) in Newly Diagnosed Malignant Glioma Patients Experiencing Fatigue Secondary to External Beam Radiation Therapy and Concurrent Temozolomide
Brief Title: Nuvigil or Placebo in Newly Diagnosed Malignant Glioma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual, Initiating Principal Investigator (PI) left Moffitt
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MCC-16233; C10953/6253 (Other: Cephalon, Inc.)
Record Dates: First submitted 2011-07-21; First posted 2011-07-25 (Estimated); Results first posted 2013-12-16 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-10

CONDITIONS: Malignant Glioma
Keywords: fatigue; external beam radiation; EBRT; radiation therapy; placebo; cognitive function; TMZ; Temozolomide
MeSH Terms: conditions — Glioma; Fatigue | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: Nuvigil® (Active Comparator): Study evaluation times correspond to standard follow-up evaluations for newly diagnosed malignant glioma patients. After 6 weeks of concurrent External Beam Radiation Therapy (EBRT) and Temozolomide (TMZ), there is typically a 4 week treatment break prior to the start of the 6 monthly cycles of TMZ. No further placebo or Nuvigil® will be given after the 6 week treatment regimen. Thus, study evaluations will occur at baseline (Week 0), immediately after completion of EBRT, TMZ, and Nuvigil® or placebo (Week 7), at the end of the 4 week washout period (Week 10), after the first 2 cycles of TMZ (Week 18), and after the 6th cycle of TMZ (Week 34).
  Interventions: Drug: Nuvigil®
- B: Placebo (Placebo Comparator): Study evaluation times correspond to standard follow-up evaluations for newly diagnosed malignant glioma patients. After 6 weeks of concurrent EBRT and TMZ, there is typically a 4 week treatment break prior to the start of the 6 monthly cycles of TMZ. No further placebo or Nuvigil® will be given after the 6 week treatment regimen. Thus, study evaluations will occur at baseline (Week 0), immediately after completion of EBRT, TMZ, and Nuvigil® or placebo (Week 7), at the end of the 4 week washout period (Week 10), after the first 2 cycles of TMZ (Week 18), and after the 6th cycle of TMZ (Week 34).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nuvigil® — Nuvigil® 150 mg/day x 42 days THEN, No More Drug
  Other Names: Armodafinil
  Arms: A: Nuvigil®
Drug: Placebo — Placebo x 42 days; THEN, No More Placebo
  Arms: B: Placebo

SUMMARY:
The purpose of this study is to determine if Nuvigil® improves fatigue experienced by people receiving external beam radiation therapy for the treatment of malignant gliomas. It is also being done to determine if Nuvigil® improves cognitive function (perception, thinking, reasoning, and remembering) and overall quality of life in people receiving external beam radiation therapy for the treatment of malignant gliomas. Another purpose of this study is to see if people who receive Nuvigil® have more or less side effects than people who receive placebo. Placebo is a substance that looks like an active drug but has no active ingredient.

DETAILED DESCRIPTION:
Study visit times will correspond with standard follow-up evaluations for the patient's malignant glioma.

Study visits will occur at baseline (Week 0); Week 7, which is when patients stop their use of study drug and their first round of external beam radiation therapy and temozolomide; and at Weeks 10, 18, and 34.

The Week 7 evaluation will include: neuropsychological exam, Psychosocial Questionnaires, and questions about the patient's medications and health.

The Week 10 and 18 evaluations will include: vital sign measurements, Karnofsky Performance status rating, neurological and neuropsychological exams, psychosocial questionnaires, an Magnetic Resonance Imaging (MRI) of the patient's brain, and questions about their medications and health.

The Week 34 evaluation will include: vital sign measurements, Karnofsky Performance status rating, neurological and neuropsychological exams, psychosocial questionnaires, and questions about the patient's medications and health.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 years or greater at study entry
* Histologic diagnosis of a supratentorial World Health Organization (WHO) grade 3 anaplastic glioma (including astrocytoma, oligodendroglioma, and mixed oligoastrocytoma) or WHO grade 4 glioblastoma which requires external beam radiation therapy (EBRT) and concurrent temozolomide (TMZ)
* Have adequate renal and liver function as evidenced by the following screening lab values: Creatinine ≤ 1.7mg/dl; Total Bilirubin ≤ 1.5mg/dl; Transaminases ≤ 4 times above the upper normal limit; Prothrombin time/international normalized ratio (PT/INR) < 1.4 for patients not on warfarin
* Adequate bone marrow functions as defined by the following lab values: Absolute neutrophil count (ANC) ≥ 1,500/mm³; Platelets ≥ 100,000 cells/mm³; Hemoglobin ≥ 10.0 gm/dL; White blood cell count (WBC) ≥ 3,000/mcL
* Karnofsky Performance Status ≥ 60%
* Recovered from the immediate neurosurgical post-operative period (e.g. for craniotomy, at least a 2 week period of time to allow for wound healing)
* Agrees to use acceptable birth control method(s). Females using steroidal contraception (oral, depot, or implantable) must agree to use an alternative or concomitant method of contraception throughout therapy as well as for one month after discontinuation of therapy.
* Agrees to avoid alcohol consumption while on therapy

Exclusion Criteria:

* Pre-existing documented traumatic brain injury
* Pre-existing dementing illness due to degenerative, cerebrovascular, or other static or progressive neurologic process
* Neurological deficit such as hemineglect or homonymous hemianopsia on baseline neurologic examination that would preclude effective participation in cognitive testing
* Intracranial space occupying lesion other than malignant glioma or benign asymptomatic meningioma
* Prior treatment with EBRT or stereotactic radiosurgery (SRS) to the brain
* Prior treatment with Nuvigil® or Provigil® within 4 weeks prior to study entry
* Leptomeningeal disease suggested clinically or by radiographic criteria
* History of left ventricular cardiac hypertrophy
* Ischemic ECG changes, chest pain, arrhythmia, or other clinically significant manifestations of mitral valve prolapse in association with central nervous system (CNS) stimulant use within the past 6 months
* Unstable angina or myocardial infarction within the past 6 months
* Premorbid or ongoing psychosis
* Currently receiving Ritalin or Tricyclic Antidepressants. Nuvigil has been demonstrated to affect the serum levels of Triazolam and Cyclosporine. Patients taking these medications will be monitored for potential dose adjustments. Other medications that are metabolized by the cytochrome P450 pathway may be potentially affected, but have not been demonstrated to do so in clinical testing. Such medications will be monitored throughout the study for possible dose adjustments.
* Patients who are experiencing significant fatigue secondary to medical or physiologic causes other than primarily from their malignant gliomas
* Pregnant, breast-feeding, or lack of willingness to use recommended birth control methods
* Patients with known hypersensitivity to modafinil, armodafinil, or its inactive ingredients
* Patients unable to understand or comply with all conditions of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Forsyth, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was Open to Accrual at Moffitt Cancer Center 12/22/2010 to 12/28/2012.
Groups:
- Active Comparator: A: Nuvigil®: Study evaluation times correspond to standard follow-up evaluations for newly diagnosed malignant glioma patients. After 6 weeks of concurrent External Beam Radiation Therapy (EBRT) and Temozolomide (TMZ), there is typically a 4 week treatment break prior to the start of the 6 monthly cycles of TMZ. No further placebo or Nuvigil® will be given after the 6 week treatment regimen. Thus, study evaluations will occur at baseline (Week 0), immediately after completion of EBRT, TMZ, and Nuvigil® or placebo (Week 7), at the end of the 4 week washout period (Week 10), after the first 2 cycles of TMZ (Week 18), and after the 6th cycle of TMZ (Week 34).
- Placebo Comparator: B: Placebo: Study evaluation times correspond to standard follow-up evaluations for newly diagnosed malignant glioma patients. After 6 weeks of concurrent EBRT and TMZ, there is typically a 4 week treatment break prior to the start of the 6 monthly cycles of TMZ. No further placebo or Nuvigil® will be given after the 6 week treatment regimen. Thus, study evaluations will occur at baseline (Week 0), immediately after completion of EBRT, TMZ, and Nuvigil® or placebo (Week 7), at the end of the 4 week washout period (Week 10), after the first 2 cycles of TMZ (Week 18), and after the 6th cycle of TMZ (Week 34).
Period: Overall Study
Arm/Group | Active Comparator: A: Nuvigil® | Placebo Comparator: B: Placebo
Started | 3 | 3
Completed | 2 | 1
Not Completed | 1 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator: A: Nuvigil® | Placebo Comparator: B: Placebo | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 1 | 2 | 3
Age Continuous [Mean (Full Range); unit: years] | 59 [48 to 66] | 65 [53 to 72] | 62 [48 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Improved Fatigue Experience After Treatment
Description: Determine if Nuvigil® improves fatigue experienced by patients receiving external beam radiation therapy for the treatment of malignant gliomas. Participants who maintained minimal, or experienced improved fatigue experience on a scale of 0 (No fatigue) - 10 (As bad as you can imagine).
Time Frame: 5 months
Population: Available, evaluable participants with minimal fatigue at baseline
Measure: Number; unit: participants
Arm/Group | Active Comparator: A: Nuvigil® | Placebo Comparator: B: Placebo
Number analyzed (Participants) | 1 | 1
participants | 0 | 0

2. Secondary Outcome: Occurrence of Improved Cognitive Performance
Description: Determine if Nuvigil® improves cognitive function of patients receiving external beam radiation therapy for the treatment of malignant gliomas. Participants who maintained average (T=50) to slightly below average (T=40 or greater) cognitive function.
Time Frame: 5 months
Population: Available, evaluable participants with average T Score range cognitive function at baseline
Measure: Number; unit: participants
Arm/Group | Active Comparator: A: Nuvigil® | Placebo Comparator: B: Placebo
Number analyzed (Participants) | 0 | 1
participants |  | 1

ADVERSE EVENTS:
Time Frame: 1 year, 9 months
Arm/Group | Active Comparator: A: Nuvigil® | Placebo Comparator: B: Placebo
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3
Other Adverse Events (participants affected / at risk) | 2/3 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Comparator: A: Nuvigil® (N=3) | Placebo Comparator: B: Placebo (N=3)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — occurred prior to taking study drug
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Comparator: A: Nuvigil® (N=3) | Placebo Comparator: B: Placebo (N=3)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Salivary duct inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0)
Fatigue (General disorders) | 2 (3) | 2 (2)
Edema limbs (General disorders) | 1 (2) | 1 (1)
Nervous system disorders - Other (Nervous system disorders) | 2 (5) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Planned accrual of 60 participants for analysis was not met. Recruitment was closed early due to slow accrual and initiating Principal Investigator (PI) leaving Moffitt.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes